CLINICAL TRIAL: NCT00403247
Title: Double-Blind Vitamin Intervention to Lower Blood Homocysteine Levels: Amino Acid and Clinical Responses in Individuals With Schizophrenia.
Brief Title: Effect of High-Dose B-Complex Vitamins on the Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04T-536
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Homocysteine; Vitamins
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Vitamin B 12; Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): vitamin capsule
  Interventions: Dietary Supplement: Capsule with folate, Vitamin B12 & pyridoxine
- B (Placebo Comparator): placebo capsule
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Capsule with folate, Vitamin B12 & pyridoxine
  Arms: A
Other: placebo — placebo capsule
  Arms: B

SUMMARY:
The purpose of this study is to determine whether individuals with schizophrenia who will take a high dose of the B-vitamins folate, B12 and pyridoxine, may experience improvement in their symptoms.

DETAILED DESCRIPTION:
Individuals with schizophrenia often experience disturbing residual symptoms, even with the best available current treatments. Homocysteine, normally found in the body, can interfere with NMDA-glutamate receptor function, and this might be responsible for some of the symptoms of schizophrenia. This double-blind protocol will have study participants who suffer from schizophrenia take either a high-dose combination of folate, B12 and pyridoxine (a combination that can lower homocysteine in the body) or placebo for three months. Clinical measures (e.g., PANSS, CGI) will be taken to determine whether those taking the vitamin combination experience clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Schizophrenia or Schizoaffective Disorder
* Ages 18-65, male or female
* Treatment regimen includes a new-generation antipsychotic (clozapine, olanzapine,risperidone, quetiapine, ziprasidone or aripiprazole)
* Stable medication for 4 weeks prior to screening visit

Exclusion Criteria:

* Diagnosis of active substance use disorder within the last month
* Already taking vitamin supplements totaling > 400 mcg folic acid per day, or regular B12 injections
* Pregnant or breastfeeding
* Seizure disorder
* Non-English speaking
* Without capacity to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
blood homocysteine levels | 12 weeks after baseline

SECONDARY OUTCOMES:
CGI (Clinical Global Improvement) | 12 weeks after baseline
CDSS (Calgary Depression Scale for Schizophrenia) | 12 weeks after baseline
WAIS-II Memory Scale (Immediate and Delayed) | 12 weeks after baseline
WAIS Digit Symbol-Coding | 12 weeks after baseline
Wisconsin Card Sorting Test | 12 weeks after baseline
WAIS-II Letter-Number Sequencing Subtest | 12 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: William M Greenberg, M.D., Principal Investigator — The Nathan Kline Institute for Psychiatric Research
Locations (1):
- The Nathan Kline Institute for Psychiatric Research, Orangeburg, New York, United States